CLINICAL TRIAL: NCT05519150
Title: Donors With Nephrolithiasis at the Time of Transplant Evaluation (DONATE). Long Term Follow-up.
Acronym: DONATE
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Muhammad Yahya Jan, Assistant Professor of Clinical Medicine, Indiana University
Other Study IDs: 15048
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Kidney Stones
Keywords: transplant
MeSH Terms: conditions — Kidney Calculi | interventions — Blood Specimen Collection; Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stone Donors: Evaluation for kidney donation > 2 years ago, had history of kidney stones or kidney stones on imaging and successfully donated a kidney
  Interventions: Diagnostic Test: low dose radiation abdomen/pelvis CT scan (stone protocol); Procedure: Blood draw; Other: 24 hour urine collection
- Denied donors: Evaluation for kidney donation > 2 years ago, had history of kidney stones or kidney stones on imaging and were declined for donation due to history of kidney stones, Litholink abnormalities or Imaging findings
  Interventions: Diagnostic Test: low dose radiation abdomen/pelvis CT scan (stone protocol); Procedure: Blood draw; Other: 24 hour urine collection
- Non-Stone Donors: Evaluation for kidney donation > 2 years ago, with no history of kidney stones, or kidney stones on Imaging and successfully donated a kidney
  Interventions: Diagnostic Test: low dose radiation abdomen/pelvis CT scan (stone protocol); Procedure: Blood draw; Other: 24 hour urine collection

INTERVENTIONS:
Diagnostic Test: low dose radiation abdomen/pelvis CT scan (stone protocol) — Kidney donors who consent will undergo a low dose radiation abdominal CT scan to identify new kidney stones in the remaining kidney. The will come to an IU Health Hospital for a low dose radiation abdomen/pelvis CT scan (stone protocol).
Procedure: Blood draw — To compare the changes changes in eGFR in evaluated kidney donors Blood will be draw by a trained phlebotomist.
Other: 24 hour urine collection — To compare the changes in metabolic kidney stone risk parameters in 24-hour urine assessments to pre-donation urine studies in evaluated kidney donors.

SUMMARY:
We believe that kidney donors with kidney stones accepted for a donation do not have an increased risk of loss of kidney function and will not be at increased risk of symptomatic kidney stone events compared to donors without a history of kidney stones.

DETAILED DESCRIPTION:
Indiana University Health center has a large nephrology and transplant service which is well versed in taking care of kidney donors with history of kidney stones. We believe that kidney donors with kidney stones accepted for a donation do not have an increased risk of loss of kidney function and will not be at increased risk of symptomatic kidney stone events compared to donors without a history of kidney stones. In this study we are contacting past kidney donors and participants with kidney stone who were declined as kidney donors. We will use blood tests, 24-hour urine tests, computed tomography (CT) scan, patient reported medical history and medical history in the patient's chart to gather data. This data will help us compare non stone donors, stone donors, and participants with kidney stone who were declined as kidney donors.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18,
* Evaluation for kidney donation > 2 years ago, with A) no history of kidney stones, or kidney stones on Imaging and successfully donated a kidney B) either had history of kidney stones or kidney stones on imaging and either i) successfully donated a kidney or ii) were declined for donation due to history of kidney stones, Litholink abnormalities or Imaging findings
* Willing to participate and sign an informed consent.

Exclusion Criteria:

* Subjects who are currently pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 90 participants who were evaluated to donate a kidney at Indiana University (IU) School of Medicine /IU Health Transplant > 2 years ago.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
changes in eGFR and urine protein to urine creatinine ratio | >2 years
  To assess the changes in eGFR and urine protein to urine creatinine ratio in kidney donors with history of kidney stones who donated a kidney 2 or more years ago. We will compare these kidney donors with the age, sex, years since donation and body mass index matched standard (non-stone) kidney donors for absolute eGFR and protein/creatinine urine ratio change, using time as a denominator by paired t-test.

SECONDARY OUTCOMES:
changes in metabolic kidney stone risk parameters in 24-hour urine assessments to pre-donation urine studies | >2 years
  To compare the changes in metabolic kidney stone risk parameters in 24-hour urine assessments to pre-donation urine studies in kidney donors with history of kidney stones compared to those who were rejected for donation due to abnormal urine studies or CT scan. We will compare pre-post 24-hour urine results for supersaturation of calcium oxalate, calcium phosphate, and uric acid (composite risks), and the individual parameters of urine volume, calcium, citrate, oxalate, uric acid and pH with paired t-test.
assess formation of new kidney stones by imaging | >2 years
  To assess formation of new kidney stones by imaging. Kidney donors who consent will undergo a low dose radiation abdominal CT scan to identify new kidney stones in the remaining kidney. We will determine the number of symptomatic, passed, and asymptomatic kidney stones on CT scan post donation as a function of time.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States